CLINICAL TRIAL: NCT07195968
Title: A Prospective, Multicenter Study: Comparative Analysis of NTG-Pd/Pa and Saline-Pd/Pa
Brief Title: Comparative Analysis of NTG-Pd/Pa and Saline-Pd/Pa (CANS)
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Miaoli General Hospital, Ministry of Health and Welfare, Taiwan (Unknown); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202507242RINB
Record Dates: First submitted 2025-09-18; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Fractional flow reserve; NTG-Pd/Pa; Saline-Pd/Pa
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cohort A: Participants will undergo NTG-Pd/Pa, saline-Pd/Pa, and FFR assessments sequentially. Saline-Pd/Pa will be tested repeatedly during the assessment.
  Interventions: Diagnostic Test: NTG-Pd/Pa measurement; Diagnostic Test: Saline-Pd/Pa measurement

INTERVENTIONS:
Diagnostic Test: NTG-Pd/Pa measurement — The coronary artery with intermediate stenosis will sequentially undergo NTG-Pd/Pa, saline-Pd/Pa, and FFR assessments. Intracoronary NTG dosage will follow the protocol based on blood pressure.
Diagnostic Test: Saline-Pd/Pa measurement — The coronary artery with intermediate stenosis will sequentially undergo NTG-Pd/Pa, saline-Pd/Pa, and FFR assessments. Ten millilitres of intracoronary saline will be given over five seconds.

SUMMARY:
The goal of this observational study is to compare the value of NTG-Pd/Pa and saline-Pd/Pa in participants with intermediate stenosis of the coronary artery. The main questions it aims to answer are:

The numerical difference between NTG-Pd/Pa and saline-Pd/Pa To compare the diagnostic performance of NTG-Pd/Pa and saline-Pd/Pa in predicting the binary result of FFR assessment?

Participants will undergo NTG-Pd/Pa, Saline-Pd/Pa, and FFR successively in the target vessel.

DETAILED DESCRIPTION:
Fractional Flow Reserve (FFR) is the gold standard for determining the functional ischemia of coronary arteries with intermediate lesions. Both intracoronary nitroglycerine (NTG) administration and saline administration induce an acute drop in trans-lesional coronary pressure. Both pressure ratios correlate well with FFR values and can reliably predict positive results in FFR assessments. The aims of this study were

1. To evaluate the numerical difference between NTG-Pd/Pa and saline-Pd/Pa.
2. To test the repeatability of saline-Pd/Pa.
3. To compare the diagnostic performance of NTG-Pd/Pa and saline-Pd/Pa in predicting the binary result of FFR assessment.

Participants will be enrolled prospectively from National Taiwan University Hospital Hsinchu Hospital, Miaoli General Hospital, and Taichung Veterans General Hospital. The coronary artery with intermediate stenosis will undergo NTG-Pd/Pa, saline-Pd/Pa, and FFR assessments sequentially. Saline-Pd/Pa will be tested repeatedly during the assessment.

ELIGIBILITY:
Inclusion Criteria:

* Participants with coronary artery with 50-90% stenosis.
* In participants who suffered from ST elevation myocardial infarction within 5 days, only the non-culprit vessel was eligible for coronary functional testing.

Exclusion Criteria:

* Systolic blood pressure is less than 90 mmHg for more than 5 minutes during examination.
* Resting heart rate is less than 50 beats per minute.
* Heart failure remains decompensated at the time of examination, such as inability to lie flat or cardiogenic shock.
* Acute onset of asthma or chronic obstructive pulmonary disease.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants referred for coronary angiography with intermediate lesions will be invited to join the registry. Enrollment sites include medical facilities in northern and central Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-17 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Absolute difference between NTG-Pd/Pa and Saline-Pd/Pa value | 3 minutes
  The absolute difference was calculated as the Saline-Pd/Pa value minus the NTG-Pd/Pa value.

SECONDARY OUTCOMES:
Diagnostic performance of NTG-Pd/Pa and Saline-Pd/Pa | 4 minutes
  To compare the diagnostic performance of NTG-Pd/Pa and saline-Pd/Pa in predicting the binary result of FFR≤0.80.
Repeatability of Saline-Pd/Pa | 2 minutes
  Saline-Pd/Pa will be measured at one-minute intervals, and the absolute differences between consecutive measurements will be analyzed.

OTHER OUTCOMES:
Target vessel failure | 3 years
  The target vessel failure included target vessel myocardial infarction, target vessel restenosis or revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Chien Boon Jong, MD, Study Chair — National Taiwan University Hospital, Hsin-Chu Hospital
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital Hsin-Chu Hospital, Hsinchu, Select
  - Miaoli General Hospital, Ministry of Health and Welfare, Miaoli
  - Taichung Veterans General Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared publicly because of ethical restrictions. The restrictions apply to the availability of these data, which were used under license for the current study, and so are not publicly available. Data are from the National Taiwan University Hospital Ethics Committee (contact via ntuhrec@ntuh.gov.tw) for researchers who meet the criteria for access to confidential data.